CLINICAL TRIAL: NCT05399212
Title: A New Natural Origin Product, Achieving More Than 80% Efficiency in Spermatogenesis in the Seminiferous Tubules. This Method Opens up Hope for Cases of Infertility Caused by the Inability of Spermatogonia to Develop Into Mature Sperm.
Brief Title: Composition for Treating Spermatogenesis and Semen Disorders / FPT-20
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trieu, Nguyen Thi, M.D. (Individual)
Collaborators: TRAN MINH DUC, MD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Therapy to spermatogenesis
Record Dates: First submitted 2022-05-21; First posted 2022-06-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Spermatogenesis and Semen Disorders
Keywords: Spermatogenesis; Male infertility; Orchitis; Mumps virus; Hypogonadism
MeSH Terms: conditions — Infertility, Male; Orchitis; Hypogonadism

STUDY DESIGN:
Intervention Model Description: The number of infertile people after recruitment was divided into 2 groups.
  * Spermatogenesis.
  * Male infertility group due to lack of sperm.
Masking Description: The number of infertile people after recruitment was divided into 2 groups.
  * Spermatogenesis.
  * Male infertility group due to lack of sperm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FPT-20 (Experimental): FPT-20 should be used regularly (>6 to 12 months) until the therapeutic purpose is achieved.
  Interventions: Drug: FPT-20

INTERVENTIONS:
Drug: FPT-20 — FPT-20 should be used regularly, the daily maintenance dose is 1 tablet once a day(>6 to 12 months) until the therapeutic purpose is achieved.

SUMMARY:
Research to develop a new, natural-derived formulation that eliminates inflammatory tissue and regenerates new tissue of the lobules, epithelium of the tubules, and connective tissue surrounding the seminiferous tubules in the testes. It restores Leydig cells and Sertoli cells' function (because the inflamed testicles were unable to perform spermatogenesis).

DETAILED DESCRIPTION:
FPT-20 has stabilized cortisol levels, maintained stable B-lymphocytes in the body, verified by quantitative tests of blood B-lymphocytes and blood cortisol, cut off the chronic inflammation chain, promoted the regeneration of the epithelium of the coiled ducts, and repairs the connective tissue surrounding the coils.

Select a type of flavonoid that has the ability to protect human body cells by destroying toxic proteins. Targeted flavonoids are selected for multiple simultaneous effects, acting as a chemotactic or physiological modifier. Many studies have shown that flavonoids can also act as cell cycle inhibitors, which can also cause cancer cell death at an early stage (at the stage of a few cells). There have been many documents demonstrating that some flavonoids have the ability to kill cancer cells, stabilize stages of cell differentiation, and improve immunity. Flavonoids present in FPT-20 protect and regenerate cells, clean up inflammatory and fibrotic cells, and facilitate the growth of germ cells.

The selected flavonoids in the preparation are also used to regenerate the epithelium in the lumen of the seminiferous tubules, ensure the perfusion of the lobules, and stabilize the spermatogenesis process.

FPT-20 is easily distributed in high concentrations in immune cells. It has natural antibacterial activity, promotes lymphocyte proliferation, and is rapidly consumed during inflammation. The effects show a prominent role in the regulation of the immune system, and there is a high degree of interaction, which requires more research to understand its mechanism, FPT-20 will not be effective in the absence of one of the components selected to participate in the test.

FPT-20 will reach its therapeutic effect after 6-12 months. After 6-12 months, an amount of progressively motile sperm was found in the semen.

According to research, FPT-20 created a homeostasis, protecting cell membranes, cutting off the cell's inflammatory chain, and preventing transcription and translation errors. The mediators regulated the protective responses in the body. Cytokines that have a beneficial effect through specific receptors, and many other unexplained processes, have altered the spermatogenesis status of the testes. The body will absorb the components in FPT-20 through the small intestine wall, this metabolism has created a significant amount of B lymphocytes to provide for the process of restoring the function of the testicles. An appropriately calculated dose of FPT-20 is provided during the treatment, using precursors, enzymes, and flavonoids available in nature to supplement and interfere with biochemical processes taking place in the body. The extracts in the preparation should be used regularly (>6 months) until the therapeutic purpose is achieved. The product has offered hope to patients who are unable to produce sperm from spermatogonia (because the process has been disrupted). Stabilize the semen pH within good limits, to produce high-quality sperm as well as to achieve efficiency into egg penetration.

ELIGIBILITY:
Inclusion Criteria:

* The selected person has evidence of spermatogenesis disorder, no sperm, and weak sperm that do not meet the standards in terms of quantity and quality.
* There are signs of orchitis.
* Accepting patients with other comorbidities such as metabolic diseases, congenital or acquired immunodeficiency, HIV/AIDS, HBV, HCV, and Tuberculosis.

Exclusion Criteria:

* Do not select patients with advanced cancer.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Carries the sex chromosome gene XY
Enrollment: 60 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Use FPT-20 drugs to increase sperm count in semen. | 180 days
  Count the number of sperm in the semen.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Thi Trieu, Dr., Study Chair — Trieu, Nguyen Thi, M.D.
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Hồ Chí Minh, Ho Chi Minh City, Vietnam